CLINICAL TRIAL: NCT04934241
Title: The Effect of Self-Acupressure on Pain and Sleep in Coronary Artery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, Zülfünaz ÖZER, PhD., Assistant Prof, Istanbul Sabahattin Zaim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 27897
Record Dates: First submitted 2021-06-15; First posted 2021-06-22 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Coronary Artery Disease
Keywords: Self-Acupressure; Sleep; Pain; Coronary Artery Patıent
MeSH Terms: conditions — Coronary Artery Disease; Pain

STUDY DESIGN:
Intervention Model Description: This study is an experimental study with pre-test and post-test control groups
Who Masked: Participant
Masking Description: Self-Acupressure and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Acupressure (Experimental): Self-Acupressure Each application to the acupressure points (HT 7, CV17,PC 6, LI4,SP 6) will be done in 2 minutes and right and left)
  Interventions: Other: Self-Acupressure
- Control group (No Intervention): Routine maintenance will be applied

INTERVENTIONS:
Other: Self-Acupressure — Acupressure is a therapy method performed with an instrument or hand, fingertip, palm, elbow, knee, thumb relaxation and wrist bands on various points representing the waist organs in order to ensure the continuation and balance of the energy in our body
  Arms: Self-Acupressure

SUMMARY:
This study will be conducted to evaluate the effect of acupressure applied to patients with coronary artery disease (CAD) on pain and sleep quality.

DETAILED DESCRIPTION:
Self-Acupressur application will improve pain and sleep quality in CAD.

ELIGIBILITY:
Inclusion Criteria:

* Not having a psychiatric diagnosis,
* To be able to communicate adequately
* Not having psychiatric problems
* Volunteering to participate in research

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-08-09 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 1. week
  The patients were asked to mark their level of pain during relaxation or activities on a 10 cm vertical or horizontal line.
  In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. VAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm
Visual Analog Scale (VAS) | 4. week
  The patients were asked to mark their level of pain during relaxation or activities on a 10 cm vertical or horizontal line.
  In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. VAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm
Pittsburgh Sleep Quality Index (PSQI) | 1. week
  The PSQI is a valid and consistent survey comprising of 19 questions to assess quality and amount of sleep and the existence of a sleep disorder and its level in the previous month. The scale was adapted into the Turkish language by Agargün et al. (1996). The scale consists of seven components that assess patients subjective sleep quality, sleep delay, use of sleeping medication and disfunction in daily activities. Each item scores in the range 0-3 points and the total score of the seven components gives the total PSQI score. The total score has a value between 0-21 and a high total score demonstrates a poor quality of sleep. A total PSQI score which is ≤5 indicates "good sleep", and a score which is >5 indicates "poor sleep"
Pittsburgh Sleep Quality Index (PSQI) | 4. week
  The PSQI is a valid and consistent survey comprising of 19 questions to assess quality and amount of sleep and the existence of a sleep disorder and its level in the previous month. The scale was adapted into the Turkish language by Agargün et al. (1996). The scale consists of seven components that assess patients subjective sleep quality, sleep delay, use of sleeping medication and disfunction in daily activities. Each item scores in the range 0-3 points and the total score of the seven components gives the total PSQI score. The total score has a value between 0-21 and a high total score demonstrates a poor quality of sleep. A total PSQI score which is ≤5 indicates "good sleep", and a score which is >5 indicates "poor sleep"

CONTACTS AND LOCATIONS:
Overall Officials: Zülfünaz ÖZER, PhD, Study Chair — Istanbul Sabahattin Zaim University
Locations (1):
- Istanbul Sabahattin Zaim University, Faculty of Health Sciences, Istanbul, Küçükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Narimani M, Ansari Jaberi A, Negahban Bonabi T, Sadeghi T. Effect of Acupressure on Pain Severity in Patients Undergoing Coronary Artery Graft: A Randomized Controlled Trial. Anesth Pain Med. 2018 Oct 20;8(5):e82920. doi: 10.5812/aapm.82920. eCollection 2018 Oct. PMID 30538941